CLINICAL TRIAL: NCT02213497
Title: Phase I Dose Escalation of Neoadjuvant Proton Beam Radiotherapy With Concurrent Chemotherapy in Locally Advanced Esophageal Cancer
Brief Title: Dose Escalation of Neoadjuvant Proton Beam Radiotherapy With Concurrent Chemotherapy in Locally Advanced Esophageal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 01214
Record Dates: First submitted 2014-08-04; First posted 2014-08-11 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Neoadjuvant; Proton Beam Radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Fluorodeoxyglucose F18; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation of Neoadjuvant Proton Radiotherapy in Esophageal Cancer (Experimental): Patients with esophageal cancer to be treated with concurrent preoperative chemoradiation with carboplatin and paclitaxel.
  Interventions: Radiation: 18F-FDG (Fluorodeoxyglucose) PET; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Radiation: 18F-FDG (Fluorodeoxyglucose) PET
Drug: Carboplatin
Drug: Paclitaxel

SUMMARY:
Patients with esophageal cancer to be treated with concurrent preoperative proton therapy along with carboplatin and paclitaxel.

DETAILED DESCRIPTION:
1. To identify the maximally tolerated radiation dose (MTD) of dose-escalated proton radiotherapy in combination with carboplatin/paclitaxel in the preoperative setting for esophageal cancer.
2. To estimate pathologic response rates by esophagectomy surgical specimens after escalated doses of chemoradiotherapy.
3. To assess the utility of circulating tumor cells and tumor vesicles as biomarkers to predict treatment response to chemoradiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of adenocarcinoma of the esophagus located distal to the carina
* Patients with AJCC 7th edition clinical stage IIB-IIIC
* Patient must be >18 years of age.
* Patients must have an ECOG Performance Status of 0-1
* Patients must be able to provide informed consent.
* Patients must be surgical candidates with adequate hematologic, renal, hepatic and pulmonary function
* serum AST and ALT < 2 times the upper limit of normal
* Patients must have bilirubin < 1.5 × normal.
* WBC > 3000/mm3, platelets > 100,000 mm3.
* Hemoglobin > 10 g/dL serum creatinine < 1.5 times the upper limit of normal
* Women of child-bearing potential as long as she agrees to use a recognized method of birth control (e.g. oral contraceptive, IUD, condoms or other barrier methods etc.). Hysterectomy or menopause must be clinically documented.

Exclusion Criteria:

* Patients with primary tumors exceeding 8 cm in length or 5 cm in width ( length should be measured by endoscopic findings, width should be measured by diagnostic CT or CT portion of PET/CT)
* Patients with primary tumors located at or above the carina
* Prior or simultaneous malignancies within the past two years (other than cutaneous squamous or basal cell carcinoma, melanoma in situ or thyroid carcinoma)
* Pregnant women, women planning to become pregnant and women that are nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-04; Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: John Plastaras, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States